CLINICAL TRIAL: NCT05104801
Title: A Phase II Study Exploring the Safety, Tolerability and Preliminary Anti-tumor Activity of Sitravatinib With or Without Tislelizumab in Patients With Unresectable or Metastatic Melanoma
Brief Title: Sitravatinib With or Without Tislelizumab in Patients With Unresectable or Metastatic Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Vice President, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-900-2002-IIT
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — sitravatinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: tislelizumab+sitravatinib (Experimental): Patients will receive sitravatinib 100 mg orally once daily in combination with tislelizumab 200 mg IV once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: sitravatinib; Drug: tislelizumab
- Arm B: sitravatinib (Experimental): Patients will receive sitravatinib 100 mg orally once daily until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: sitravatinib

INTERVENTIONS:
Drug: sitravatinib — sitravatinib 100mg QD PO
Drug: tislelizumab — tislelizumab 200mg Q3W IV
  Arms: Arm A: tislelizumab+sitravatinib

SUMMARY:
In 2014, an estimated 7,000 patients were diagnosed of melanoma in China. It is growing at an annual rate of 3%-5% and approximately 20,000 new cases are reported each year recently.To date, CFDA only approved dacarbazine as first line chemotherapy and anti-PD-1 antibody monotherapy as second line. There is no standard of care after chemotherapy and anti-PD-1.

DETAILED DESCRIPTION:
This is an open-label, randomized, single center phase 2 study evaluating the efficacy and safety of sitravatinib in combination with tislelizumab for Chinese patients with unresectable or metastatic melanoma after disease progression from prior anti-PD-1 antibody and chemotherapy. The first 20 patients will be randomized in a 1:1 ratio to receive either sitravatinib plus tislelizumab (Arm A) or sitravatinb monotherapy (Arm B). After the completion of initial 20 patients, additional patients will be recruited until 24 efficacy evaluable patients achieved in Arm A

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the Schedule of Assessments
2. Age ≥ 18 years on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place)
3. Disease progression from prior chemotherapy and anti-PD-(L)1 therapy (including sequential or combined therapy, regardless of the order)
4. No antiPD-1/PD-L1 related toxicity during the prior treatment
5. Have not received other immunotherapy, including but not limited to anti-OX40, anti-TIGIT and anti-CD137, etc.
6. BRAF wild-type patients, or patients with BRAF mutations who are not suitable or refused to receive targeted therapy with BRAF inhibitors and/or MEK inhibitors
7. Have not been exposed to small molecule targeted drugs with anti-angiogenesis effect, or VEGFR TKI drugs
8. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
9. Adequate hematologic and end-organ function
10. Have not received radiotherapy, endocrine therapy, molecular targeted therapy, or surgery within 2 weeks before the start of the study, and have recovered from the acute toxicity of the previous treatment
11. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and ≥ 120 days after the last dose of study drugs and have a negative serum pregnancy test ≤ 7 days of first dose of study drugs

Exclusion Criteria:

1. Ocular melanoma
2. known NRAS mutations
3. Active leptomeningeal disease or brain metastases that are not well controlled.
4. History of active autoimmune disease
5. Any active malignancy ≤ 2 years
6. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before first dose of study drugs
7. History of interstitial lung disease, noninfectious pneumonitis or uncontrolled diseases, including pulmonary fibrosis, acute lung diseases, etc.
8. Severe chronic or active infections (including tuberculosis infection, etc.) requiring systemic antibacterial, antifungal or antiviral therapy, within 14 days prior to first dose of study drugs
9. Known history of HIV infection
10. Any major surgical procedure requiring general anesthesia ≤ 28 days before first dose of study drugs
11. Prior allogeneic stem cell transplantation or organ transplantation
12. Hypersensitivity to tislelizumab or sitravatinib, to any ingredient in the formulation, or to any component of the container
13. Bleeding or thrombotic disorders or use of anticoagulants such as warfarin or similar agents requiring therapeutic INR monitoring within 6 months before first dose of study drugs
14. Concurrent participation in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) in Arm A | 12 months
  defined as the proportion of participants with partial response or complete response as determined by the investigators based on RECIST v1.1

SECONDARY OUTCOMES:
Overall response rate (ORR) in Arm B | 12 months
  defined as the proportion of participants with partial response or complete response as determined by the investigators based on RECIST v1.1
Disease control rate (DCR) in Arm A and B | 12 months
  defined as the proportion of participants whose best overall response (BOR) is complete response, partial response or stable disease as determined by investigators based on RECIST v1.1
Progression-free survival (PFS) in Arm A and B | 12 months
  defined as the time from randomization to the first occurrence of disease progression as determined by the investigator based on RECIST v1.1, or death from any cause, whichever occurs first
Incidence of Treatment-Emergent Adverse Events | 12 months
  According to National Cancer Institute Common Terminology Criteria for Adverse Events V5.0(CTCAE V5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No